CLINICAL TRIAL: NCT04188665
Title: Using Maackia Amurensis Seed Lectin to Target the Podoplanin Receptor As a Functionally Relevant Biomarker to Inhibit the Growth of Oral Squamous Cell Carcinoma and Precancerous Lesions
Brief Title: Using MASL to Combat Oral Cancer
Status: Active, not recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Rowan University (Other)
Collaborators: Rutgers University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Pro2019000548
Record Dates: First submitted 2019-11-19; First posted 2019-12-06 (Actual); Last update posted 2025-01-13 (Actual); Status verified 2025-01

CONDITIONS: Squamous Cell Carcinoma of Head and Neck
Keywords: maackia amurensis; podoplanin; pdpn; lectin; oral squamous cell carcinoma
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- MASL treated (Experimental): Patients treated with lozenge containing MASL
  Interventions: Drug: MASL
- Placebo treated (Placebo Comparator): Patients treated with lozenge without MASL
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: MASL — Patients treated with MASL lozenge
  Other Names: Maackia amurensis seed lectin
  Arms: MASL treated
Other: Placebo — Patients treated with placebo lozenge
  Arms: Placebo treated

SUMMARY:
This project will evaluate the expression of a receptor called podoplanin (PDPN) in cells from oral cancers and precancerous lesions. We will also determine how sensitive oral cancer cells are to a potential drug called Maackia amurensis seed lectin (MASL).

ELIGIBILITY:
Inclusion Criteria:

1. Males and females of at least 18 years of age who are able to give consent.
2. Smokers and non-smokers.
3. Persons with white or red spots and/or lesions suspected or found to be oral cancer or precancer on the inner surface of the mouth.
4. Oral lesions will be classified as OSCC or leukoplakia including, proliferative verrucous leukoplakia, conventional erythroplakia, suspect oral papillomas, or oral lichen planus. Only patients with such histologically confirmed diagnoses will be considered for inclusion.
5. patients will be considered for inclusion at any stage of disease progression.
6. Patients will be considered for inclusion if a subsequent biopsy or surgical resection are planned as part of their best care treatment.
7. Patients will have an Eastern Cooperative Oncology Group performance status of 0 or 1.
8. Patients will display normal organ function as evidenced by standard laboratory blood tests including liver enzymes and creatine.
9. Patients will not present evidence of comorbidities including ongoing or active infection, unstable illness, or medical conditions.

Exclusion Criteria:

1. Patients with cognitive impairments and cannot consent for themselves.
2. Patients with language/hearing impairments.
3. Use of a topical steroid product within the last 2 weeks.
4. Pregnant women (to avoid any potential risk to the fetus) to be confirmed by standard blood or urine tests according to best care practice.
5. Patients who are breastfeeding.
6. Abstinence or use of adequate contraception will be required for women of childbearing potential and men of reproductive potential.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2021-01-29 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Pre-treatment OSCC morphology and PDPN expression | 1 day to 4 weeks.
  Measure morphology and podoplanin (PDPN) expression by immunohistochemistry of cells included in initial biopsies of oral lesions in comparison to normal oral squamous epithelial cells (OSCCs). We will select patients with lesions that express robust levels of PDPN and notable dysplasia for inclusion in the study.

SECONDARY OUTCOMES:
Post-treatment OSCC morphology and PDPN expression | 1 day to 4 weeks.
  Evaluate and compare the PDPN expression and morphology of cells from included in resected oral lesions from patients treated with the experimental compound MASL or placebo. We will measure if MASL treatment decreases PDPN expression and normalizes morphology of OSCC cells on a defined scale of pathological examination by immunohistochemistry.

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - New Jersey Medical School, Newark, New Jersey
  - Rutgers School for Dental Medicine, Newark, New Jersey
  - University Hospital, Newark, New Jersey
  - Rowan University, Stratford, New Jersey